CLINICAL TRIAL: NCT01716572
Title: Erythromycin Versus Gastric Lavage to Improve Quality of Endoscopic Examination in Patients With Upper Gastrointestinal Bleeding. A Prospective Randomized Trial.
Brief Title: Erythromycin Versus Gastric Lavage to Improve Quality of Endoscopy in Patients With Upper Gastrointestinal Bleeding
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Principal Investigator, Dr Antonio Soriano Izquierdo, Physician Doctor, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERITRO2011
Record Dates: First submitted 2012-06-28; First posted 2012-10-30 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Gastrointestinal Hemorrhage; Hematemesis
Keywords: Upper gastrointestinal bleeding; Endoscopy; Erythromycin; Gastric lavage
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hematemesis | interventions — Erythromycin; Gastric Lavage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- gastric lavage (Active Comparator): gastric lavage by nasogastric tube with 1 liter saline before the endoscopy
  Interventions: Procedure: gastric lavage
- erythromycin (Active Comparator): administration of 250mgr of erythromycin before the endoscopy
  Interventions: Drug: Erythromycin

INTERVENTIONS:
Drug: Erythromycin — Intravenous 250 mg of erythromycin, single-dose, 30 minutes before the endoscopy
  Other Names: Pantomicina Intravenosa
  Arms: erythromycin
Procedure: gastric lavage — gastric lavage by nasogastric tube with 1 liter of saline before the endoscopy
  Arms: gastric lavage

SUMMARY:
The researchers will investigate whether erythromycin infusion is better than gastric lavage prior to emergency endoscopy to improve the quality of examination in patients with upper gastrointestinal bleeding.

DETAILED DESCRIPTION:
The researchers will investigate whether erythromycin infusion is better than gastric lavage prior to emergency endoscopy to improve the quality of examination in patients with upper gastrointestinal bleeding.

One hundred and twenty-two patients admitted within 12 hours after hematemesis will be randomly assigned to receive erythromycin infusion or gastric lavage by nasogastric tube prior to emergency endoscopy. The endoscopic procedures will be recorded on Digital Video Disc (DVD). Two endoscopists blinded to the cleansing strategy will assess the quality of examination of the upper gastrointestinal tract by using scales designed by Frossard and Avgerinos .

Secondary endpoints will be the need for a second-look endoscopy, the mean number of blood units transfused, the need of surgery or arteriography, and the mean duration of hospitalization

ELIGIBILITY:
Inclusion Criteria:

* recent hematemesis (<12 hours)

Exclusion Criteria:

* macrolides allergy
* pregnancy or lactation
* treatment with terfenadine, astemizole or cyclosporine
* prior gastrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Visual quality of endoscopy | The endoscopy will be recorded and subsequently it will be evaluated by two endoscopists unaware of the cleaning strategy. The recording's evaluation will be made within the first 30 days after endoscopy
  To assess the visual quality of endoscopy the investigators will use the Avgerinos' score modified by Frossard (Gastroenterology 2002;123:17-23). An score from 0 to 2(0 worst vision, where < 25% of the surface was visible. 1, 25-75% visible and 2 >75% visible) was derived from analysis of each area (fundus, body, antrum and bulbus). A score of 6 or greater is considered as a clear stomach, and a score of 5 or lower was considered as a full stomach.

SECONDARY OUTCOMES:
need for a second-look endoscopy | within the first 30 days after endoscopy
  To assess the need of a second-look endoscopy due to a full stomach during the first endoscopy or due to rebleeding
need of blood transfusion | within 30 days after endoscopy
number of adverse events as a measure of safety and tolerability | within the first 30 days after endoscopy
length of hospitalisation | within the first 30 days after endoscopy
length of endoscopic procedure | within the first 30 days after endoscopy
need for arteriography or surgery | within the first 30 days after endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Soriano, M D, Ph D, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Frossard JL, Spahr L, Queneau PE, Giostra E, Burckhardt B, Ory G, De Saussure P, Armenian B, De Peyer R, Hadengue A. Erythromycin intravenous bolus infusion in acute upper gastrointestinal bleeding: a randomized, controlled, double-blind trial. Gastroenterology. 2002 Jul;123(1):17-23. doi: 10.1053/gast.2002.34230. PMID 12105828
- [Background] Coffin B, Pocard M, Panis Y, Riche F, Laine MJ, Bitoun A, Lemann M, Bouhnik Y, Valleur P; Groupe des endoscopistes de garde a l'AP-HP. Erythromycin improves the quality of EGD in patients with acute upper GI bleeding: a randomized controlled study. Gastrointest Endosc. 2002 Aug;56(2):174-9. doi: 10.1016/s0016-5107(02)70174-0. PMID 12145593
- [Background] Carbonell N, Pauwels A, Serfaty L, Boelle PY, Becquemont L, Poupon R. Erythromycin infusion prior to endoscopy for acute upper gastrointestinal bleeding: a randomized, controlled, double-blind trial. Am J Gastroenterol. 2006 Jun;101(6):1211-5. doi: 10.1111/j.1572-0241.2006.00582.x. PMID 16771939
- [Background] Pateron D, Vicaut E, Debuc E, Sahraoui K, Carbonell N, Bobbia X, Thabut D, Adnet F, Nahon P, Amathieu R, Aout M, Javaud N, Ray P, Trinchet JC; HDUPE Collaborative Study Group. Erythromycin infusion or gastric lavage for upper gastrointestinal bleeding: a multicenter randomized controlled trial. Ann Emerg Med. 2011 Jun;57(6):582-9. doi: 10.1016/j.annemergmed.2011.01.001. Epub 2011 Feb 17. PMID 21333385
- [Background] Barkun AN, Bardou M, Martel M, Gralnek IM, Sung JJ. Prokinetics in acute upper GI bleeding: a meta-analysis. Gastrointest Endosc. 2010 Dec;72(6):1138-45. doi: 10.1016/j.gie.2010.08.011. PMID 20970794
- [Background] Winstead NS, Wilcox CM. Erythromycin prior to endoscopy for acute upper gastrointestinal haemorrhage: a cost-effectiveness analysis. Aliment Pharmacol Ther. 2007 Nov 15;26(10):1371-7. doi: 10.1111/j.1365-2036.2007.03516.x. Epub 2007 Sep 10. PMID 17848180
- [Background] Barkun AN, Bardou M, Kuipers EJ, Sung J, Hunt RH, Martel M, Sinclair P; International Consensus Upper Gastrointestinal Bleeding Conference Group. International consensus recommendations on the management of patients with nonvariceal upper gastrointestinal bleeding. Ann Intern Med. 2010 Jan 19;152(2):101-13. doi: 10.7326/0003-4819-152-2-201001190-00009. PMID 20083829